CLINICAL TRIAL: NCT02176564
Title: COPD, Inhaled Bronchodilators Association, and Quality of Life
Brief Title: Inhaled Bronchodilator Association and Quality of Life in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1012.40
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Chronic obstructive pulmonary disease: Patients with COPD treated with inhaled bronchodilators
  Interventions: Drug: inhaled bronchodilator

INTERVENTIONS:
Drug: inhaled bronchodilator

SUMMARY:
A pharmaco-epidemiological, observational study that aimed at assessing in a prospective manner the evolution of Quality of Life (QOL) in chronic obstructive pulmonary disease (COPD) patients treated with inhaled bronchodilators

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD confirmed by Pulmonary Function Test (PFTs)
* Recent treatment with a free or fixed association of inhaled bronchodilators

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with COPD
Sampling Method: Non-Probability Sample
Enrollment: 2639 (Actual)
Dates: Start 1999-06; Primary Completion 2000-10 (Actual)

PRIMARY OUTCOMES:
Assessment of health-related quality of life (Short-Form Health Survey) | 4 months